CLINICAL TRIAL: NCT06322472
Title: The Relationship Between Phonological Awareness Skills and Home Environment Literacy in Cochlear Implant Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Büşra AKSU, Research Assistant, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 138956
Record Dates: First submitted 2024-02-19; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cochlear Implants; Child Language; Literacy; Phonological (Speech) Disorder
Keywords: cochlear implant; home environment; early literacy; phonological awareness; pediatri
MeSH Terms: conditions — Literacy; Articulation Disorders

STUDY DESIGN:
Intervention Model Description: Descriptive research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 23 children with cochlear implants (Experimental): The children with cochlear implants was applied The Early Childhood Phonological Sensitivity Scale and The Turkish Early Language Development Test.
  Interventions: Other: The Turkish Early Language Development Test (TEDIL); Other: The Early Childhood Phonological Sensitivity Scale (PASECP)
- 23 parents (Other): Demographic Questionaries, Family Literacy Scale and ELHES were applied to the families of the participants
  Interventions: Other: The Family Literacy Scale; Other: The Early Literacy Home Environment Scale (ELHES); Other: Demographic Questionaries

INTERVENTIONS:
Other: The Turkish Early Language Development Test (TEDIL) — The Turkish Early Language Development Test (TEDIL) is a test that measures the receptive and expressive language skills of children between the ages of 2 and 7 years and 11 months.
  Arms: 23 children with cochlear implants
Other: The Family Literacy Scale — The Family Literacy Scale, which is a reliable and valid measurement scale, was developed by Kılıç, Doğan, and Özden (Kılıç, Doğan, and Özden 2017). The items of the scale consist of questions about parental literacy, child literacy, and early literacy. Parental Literacy Scale to identify and analyse situations such as the use of literacy skills, role modelling for children, performing simple literacy activities at home, on the street, etc. and generally helping children to learn to read and write.
  Arms: 23 parents
Other: The Early Childhood Phonological Sensitivity Scale (PASECP) — The Early Childhood Phonological Sensitivity Scale (PASECP), developed by Sarı and Aktan Acar (2013), measures the phonological awareness of children aged 60-72 months (Sari and Aktan Acar 2013).
  Arms: 23 children with cochlear implants
Other: The Early Literacy Home Environment Scale (ELHES) — The Early Literacy Home Environment Scale (ELHES) developed by Karaahmetoğlu and Turan is a reliable and valid questionnaire for assessing the early literacy home environment of families with children aged 0-6 years (Karaahmetoğlu and Turan 2020)
  Arms: 23 parents
Other: Demographic Questionaries — The demographic survey was prepared by the researchers. The demographic survey includes questions about educational status and family's socio-economic status.
  Arms: 23 parents

SUMMARY:
The aim was to examine the relationship between home literacy of parents whose has children who use cohlear implant and family demographic characteristics and phonological awareness skills of children with cochlear implant.

DETAILED DESCRIPTION:
This study was designed to determine the relationship between home literacy of parents whose has children who use cohlear implant and family demographic characteristics and phonological awareness skills of children with cochlear implant.To collect data from the parents, "Demographic Questionary" which is prepared by the researchers, "Early Literacy Home Environment Scale (ELHES)" (Karaahmetoğlu & Turan, 2017), and "Family Literacy Scale" (Kılıç, Doğan & Özden, 2017) were used in the study. To collect data from the children with cochlear implant users, "The Turkish Early Language Development Test (TEDİL) " (Topbaş & Güven, 2013), and "The Early Childhood Phonological Sensitivity Scale (PASECP)" (Sarı & Acar, 2013) were used in the study.

This study was carried out with follow-up patients in the Audiology, Language and Speech Disorders Clinic of xxx University - Medical Faculty, Department of Otorhinolaryngology. The study was performed with the approval of Ethics Committee, and written informed consent was obtained from all patient families (138955/ July 2021). There are 23 cochlear implant users and, 23 their family. Children ranging in age from 5 to 7 who also have 5-6 years old language skills without any neurological problems were included in the study.

SPSS 25.0 (IBM) was used program for statistical analysis. The differences of the numerical measurements used in the research according to the binary demographic categories were analyzed with the Mann Whitney U test, and the analysis of the differences according to the multiple categories was analyzed with the Kruskal Wallis H test. The significance level (α=0.05) was used.

ELIGIBILITY:
Inclusion Criteria:

* language skills were between 60 and 72 months; not enrolled in primary school; regular use of unilateral or bilateral cochlear implants;regular training in an auditory rehabilitation center

Exclusion Criteria:

* The study excluded individuals who did not meet the inclusion criteria for the control and study groups.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
The data the Early Childhood Phonological Sensitivity Scale (PASECP) from children with cochlear implants | 3 months
  The Early Childhood Phonological Sensitivity Scale (PASECP) which was developed by Sarı and Aktan Acar (2013) measure phonological awareness of children aged 60-72 months. The test contains eight sub-dimensions, and total of 78 items. 1 point is taken for each correct answer. The sub-dimensions of the scale are recognizing rhyme, beginning sound detection, the generating new words related to the desired phoneme, grouping words starting with the same sound within a group of words, blending phonemes, segmenting word into its syllables, omitting a word in a compound and of alphabet knowledge. The scale was used to measure the phonological awareness skills of children with cochlear implants in the study.
The data Family Literacy Scale from parents | 1 months
  The Family Literacy Scale which a reliable and valid measurement scale was developed by Kılıç, Doğan, and Özden in 2017. The question items of the scale consist about parental literacy, child literacy, and early literacy. Parental Literacy Scale to identify and analyze situations such as using literacy skills, role modeling for children, performing simple literacy activities at home, on the street, etc., and generally helping children learn how to read and write. The questions were 32 items and rated on a five-point Likert scale. (Always=5 point, Often=4 points, Sometimes=3 points, Rarely=2 points, and Never=1 point). The higher scores on the scale indicate to increased parent literacy level. This scale used to determine the literacy status of families in this study.
The data Early Literacy Home Environment Scale (ELVES) from parents | 2 weeks
  The Early Literacy Home Environment Scale (ELHES) is a scale reliable and valid questionnaire for assessing the early literacy home environments of families with children 0-6 years of age. The scale is four-point Likert. The total score is obtained by summing all the items (the lowest score is 8, and the highest score is 32). The scale of home early literacy environment range from 8 to 32; 8-15 is "insufficient", 16-23 "medium", 24-32 "sufficient". It was used to evaluate the early literacy opportunities provided by families for children with using cochlear implants in the home environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ching TY, Cupples L. Phonological Awareness at 5 years of age in Children who use Hearing Aids or Cochlear Implants. Perspect Hear Hear Disord Child. 2015 Sep;25(2):48-59. doi: 10.1044/hhdc25.2.48. PMID 26929789
- [Background] Ahmed, Eman, Ahmed Elmesalamy, Fekry Mohamed, Hassan El-Ater, Mohamed Fekry, and El-Ater Hassan. 2022. "The Role of the Home Literacy Environment and Parent Education in Effecting the Developmental Differences of Phonological Awareness During Early Child Hood." American Journal of Applied Psychology 11 (1): 36.
- [Background] Bell, Nicola, Anthony J. Angwin, Wayne J. Wilson, and Wendy L. Arnott. 2022. "Literacy Development in Children with Cochlear Implants: A Narrative Review." Australian Journal of Learning Difficulties 27 (1): 115-34.
- [Background] Ebert S, Lehrl S, Weinert S. Differential Effects of the Home Language and Literacy Environment on Child Language and Theory of Mind and Their Relation to Socioeconomic Background. Front Psychol. 2020 Oct 29;11:555654. doi: 10.3389/fpsyg.2020.555654. eCollection 2020. PMID 33192809
- [Background] DesJardin JL, Ambrose SE, Eisenberg LS. Literacy skills in children with cochlear implants: the importance of early oral language and joint storybook reading. J Deaf Stud Deaf Educ. 2009 Winter;14(1):22-43. doi: 10.1093/deafed/enn011. Epub 2008 Apr 15. PMID 18417463
- [Background] Eyalati N, Jafari Z, Ashayeri H, Salehi M, Kamali M. Effects of parental education level and economic status on the needs of families of hearing-impaired children in the aural rehabilitation program. Iran J Otorhinolaryngol. 2013 Winter;25(70):41-8. PMID 24303418
- [Background] Hassunah-Arafat, Safieh Muhamad, Dorit Aram, and Ofra Korat. 2021. "Early Literacy in Arabic: The Role of SES, Home Literacy Environment, Mothers' Early Literacy Beliefs and Estimation of Their Children's Literacy Skills." Reading and Writing 34 (10): 2603-25.
- [Background] Incognito, Oriana, and Giuliana Pinto. 2021. "Longitudinal Effects of Family and School Context on the Development on Emergent Literacy Skills in Preschoolers." Current Psychology.
- [Background] Ingvalson EM, Grieco-Calub TM, Perry LK, VanDam M. Rethinking Emergent Literacy in Children With Hearing Loss. Front Psychol. 2020 Jan 31;11:39. doi: 10.3389/fpsyg.2020.00039. eCollection 2020. PMID 32082217
- [Background] Kim, Sojung, Haesung Im, and Kyong Ah Kwon. 2015. "The Role of Home Literacy Environment in Toddlerhood in Development of Vocabulary and Decoding Skills." Child and Youth Care Forum 44 (6): 835-52.
- [Background] Liu, Cuina, George K. Georgiou, and George Manolitsis. 2018. "Modeling the Relationships of Parents' Expectations, Family's SES, and Home Literacy Environment with Emergent Literacy Skills and Word Reading in Chinese." Early Childhood Research Quarterly 43: 1-10.
- [Background] Luo, Rufan, Amy Pace, Dani Levine, Aquiles Iglesias, Jill de Villiers, Roberta Michnick Golinkoff, Mary Sweig Wilson, and Kathy Hirsh-Pasek. 2021. "Home Literacy Environment and Existing Knowledge Mediate the Link between Socioeconomic Status and Language Learning Skills in Dual Language Learners." Early Childhood Research Quarterly 55: 1-14.
- [Background] Ngorosho, Damaris, and Ulla Lahtinen. 2010. "The Role of the Home Environment in Phonological Awareness and Reading and Writing Ability in Tanzanian Primary Schoolchildren." Education Inquiry 1 (3): 211-34.
- [Background] Pluijm, M Van Der, A Van Gelderen, and J Kessels. 2019. "Activities and Strategies for Parents With Less Education to Promote the Oral Language Development of Their Children: A Review of Empirical Interventions." School Community Journal 29 (1): 317-62.
- [Background] Riser, Quentin H., Heather L. Rouse, Ji Young Choi, and Seulki Ku. 2020. "The Contribution of Home Literacy Context to Preschool Academic Competencies for American Indian and Alaska Native Children." Child and Youth Care Forum 49 (2): 303-23. https://doi.org/10.1007/s10566-019-09529-1.
- [Background] Slicker, Gerilyn, Christina A. Barbieri, Zachary K. Collier, and Jason T. Hustedt. 2021. "Parental Involvement during the Kindergarten Transition and Children's Early Reading and Mathematics Skills." Early Childhood Research Quarterly 55: 363-76.
- [Background] Soleymani Z, Mahmoodabadi N, Nouri MM. Language skills and phonological awareness in children with cochlear implants and normal hearing. Int J Pediatr Otorhinolaryngol. 2016 Apr;83:16-21. doi: 10.1016/j.ijporl.2016.01.013. Epub 2016 Jan 25. PMID 26968046
- [Background] Su M, Li P, Zhou W, Shu H. Effects of socioeconomic status in predicting reading outcomes for children: The mediation of spoken language network. Brain Cogn. 2021 Feb;147:105655. doi: 10.1016/j.bandc.2020.105655. Epub 2020 Nov 27. PMID 33249385
- [Background] Su, Mengmeng, Hugo Peyre, Shuang Song, Catherine McBride, Twila Tardif, Hong Li, Yuping Zhang, et al. 2017. "The Influence of Early Linguistic Skills and Family Factors on Literacy Acquisition in Chinese Children: Follow-up from Age 3 to Age 11." Learning and Instruction 49: 54-63. https://doi.org/10.1016/j.learninstruc.2016.12.003.
- [Background] Turan, F., and G. Akoğlu. 2014. "Home Literacy Environment and Phonological Awareness Skills in Preschool Children | Okul Öncesi Dönemde Ev Okuryazarlık Ortamı ve Fonolojik Farkındalık Becerileri." Hacettepe Egitim Dergisi 29 (3): 153-66.
- [Background] Wang Y, Liu L, Zhang Y, Wei C, Xin T, He Q, Hou X, Liu Y. The Neural Processing of Vocal Emotion After Hearing Reconstruction in Prelingual Deaf Children: A Functional Near-Infrared Spectroscopy Brain Imaging Study. Front Neurosci. 2021 Jul 28;15:705741. doi: 10.3389/fnins.2021.705741. eCollection 2021. PMID 34393716
- [Background] Wilcox, M. Jeanne, Shelley Gray, and Mark Reiser. 2020. "Preschoolers with Developmental Speech and/or Language Impairment: Efficacy of the Teaching Early Literacy and Language (TELL) Curriculum." Early Childhood Research Quarterly 51: 124-43. https://doi.org/10.1016/j.ecresq.2019.10.005.